CLINICAL TRIAL: NCT04401007
Title: A Volunteer Study to Determine the Anesthetic and Analgesic Effect of the Erector Spinae Plane (ESP) Block
Brief Title: Erector Spinae Plane (ESP) Block Volunteer Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 19-5863.0
Record Dates: First submitted 2020-05-11; First posted 2020-05-26 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia | interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: There will be 2 study subgroups based on the vertebral level at which the ESP block is administered: (1) Volunteer subjects in subgroup TP4 will receive the ESP block injection at the T4 transverse process (TP4) level. Injection at the TP4 level will allow us to evaluate the anesthetic effect on the chest wall. (2) Volunteers in subgroup TP8 will receive the ESP block injection at the T8 transverse process (TP8) level. Injection at the TP8 level will allow us to evaluate the anesthetic effect on the abdominal wall.
  The first 12 volunteer subjects recruited will receive ESP blocks at the TP4 level and the subsequent 12 subjects will receive ESP blocks at the TP8 level.
Who Masked: Participant, Investigator
Masking Description: Two different local anesthetic volumes will be investigated: 20 mL (300 mg lidocaine) at one study visit and 30 mL (450 mg lidocaine) at the other study visit. Volunteers will be randomized to one of two intervention groups: (1) Group 20/30: A unilateral ESP block with 20 mL of local anesthetic at the first visit, and 30 mL of local anesthetic at the second visit; or (2) Group 30/20: a unilateral ESP block with 30 mL of 1.5% lidocaine with 1/200,000 epinephrine at the first visit, and 20 mL of the same local anesthetic solution at the second visit. Randomization of subjects to either Group 20/30 or Group 30/20 will be done using computer software and only the study investigator performing the ESP block will be aware of the study allocation. Volunteer subjects and the study investigators responsible for serial neurologic and other outcome assessments after injection will be blinded to the volume of local anesthetic injected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 20/30 (Experimental): Two different local anesthetic volumes will be investigated: 20 mL of 1.5% lidocaine (300 mg lidocaine) at one study visit and 30 mL of 1.5% lidocaine (450 mg lidocaine) at the other study visit. Volunteers will be randomized to one of two intervention groups: (1) Group 20/30: A unilateral ESP block with 20 mL of local anesthetic at the first visit, and 30 mL of local anesthetic at the second visit
  Interventions: Other: Erector Spinae Plane Block with 1.5% lidocaine
- Group 30/20 (Experimental): (2) Group 30/20: a unilateral ESP block with 30 mL of 1.5% lidocaine with 1/200,000 epinephrine at the first visit, and 20 mL of the same local anesthetic solution at the second visit. This crossover design allows subjects to serve as their own control.
  Interventions: Other: Erector Spinae Plane Block with 1.5% lidocaine

INTERVENTIONS:
Other: Erector Spinae Plane Block with 1.5% lidocaine — Erector spinae plane (ESP) block is a new regional nerve block technique that involves a percutaneous injection of local anesthetic as a bolus through a needle or catheter into the fascial plane between the erector spinae muscle and the transverse processes in the upper or mid back.

SUMMARY:
Although erector spinae plane (ESP) block reportedly provides postoperative pain relieve, controversy remains regarding the accuracy and consistency of analgesic success following ESP block. The goal of this study is to determine the extent and duration of clinical neural blockade following an ESP injection with different local anesthetic doses.

Methods Twenty four healthy volunteers will be recruited, and each subject will make 2 separate visits to the study centre to undergo intervention and assessment. The 2 study visits will be separated by an interval of at least 2 weeks to ensure complete washout of any residual effects and a return to baseline status.

At each study visit, the subject will receive a unilateral ESP block with 1.5% lidocaine and 5 mcg/mL epinephrine. Two different local anesthetic volumes will be investigated: 20 mL (300 mg lidocaine) at one study visit and 30 mL (450 mg lidocaine) at the other study visit. Volunteers will be randomized to one of two intervention groups: (1) Group 20/30: A unilateral ESP block with 20 mL of local anesthetic at the first visit, and 30 mL of local anesthetic at the second visit; or (2) Group 30/20: a unilateral ESP block with 30 mL of 1.5% lidocaine with 1/200,000 epinephrine at the first visit, and 20 mL of the same local anesthetic solution at the second visit.

There will be 2 study subgroups based on the vertebral level at which the ESP block is administered: (1) Volunteer subjects in subgroup TP4 will receive the ESP block injection at the T4 transverse process (TP4) level in order to evaluate the anesthetic effect on the chest wall. (2) Volunteers in subgroup TP8 will receive the ESP block injection at the T8 transverse process (TP8) level in order to evaluate the anesthetic effect on the abdominal wall. The first 10 volunteer subjects recruited will receive ESP blocks at the TP4 level and the subsequent 10 subjects will receive ESP blocks at the TP8 level.

DETAILED DESCRIPTION:
Erector spinae plane (ESP) block is a new regional nerve block technique that involves a percutaneous injection of local anesthetic as a bolus through a needle or catheter into the fascial plane between the erector spinae muscle and the transverse processes in the upper or mid back. Injection at the level of the T4-5 transverse process is indicated for chest wall pain relief while injection at the T8-9 level is for abdominal wall pain control. This block aims to relieve postoperative pain but is not intended to provide anesthetic blockade for surgery. Preliminary case reports and some randomized controlled trials show encouraging analgesic effect of ESP block for breast surgery, rib fracture, thoracotomy, sternotomy, epigastric hernia repair, open abdominal surgery, laparoscopic abdominal surgery, radical retropubic prostatectomy and hip arthroplasty. Although effective, controversy remains regarding the accuracy and consistency of analgesic success following ESP block.

Currently, it is unclear whether block inconsistency is due to improper injection technique or the mechanism of action. Presumably, local anesthetic following an ESP block injection will find its way antero-medially through the costotransverse foramen and / or inter transverse ligaments to enter the thoracic paravertebral space or epidural space to block the ventral rami of the thoracic spinal nerves. It may also spread laterally to reach the neighbouring intercostal nerves.

At this time, it is unclear whether cadaver injection studies showing dye spread to these anatomical spaces can fully explain the observed clinical neural blockade. Also a number of cadaver studies show inconsistent and conflicting dye spread results, i.e., failure to reach the thoracic paravertebral space. Although some suggest that an ESP block also provides sympathetic blockade thus may provide visceral pain relief, no study has evaluated the validity of such a claim or the extent of sympathetic blockade.

The mechanisms of action for an ESP block are currently unclear. Although most case reports describe analgesic effects of ESP block for anterior chest and abdominal surgery presumably as a result of blockade of the ventral rami of the spinal nerves in the thoracic paravertebral spaces, it is more likely that local anesthetic injected in the ESP will reliably anesthetize the dorsal rami traversing the erector spinae muscle in the back. This is supported by preliminary clinical analgesic success of ESP block for thoracic spine surgery and lumbar spine surgery. The consistency of blocking the ventral and dorsal rami following an ESP block injection is unknown at this time.

Investigators' clinical experience further confirms that an ESP injection provides variable analgesic results and an objective sign of sensory anesthesia to pinprick or ice is not consistently evident. Currently no study has examined the optimal technique of ESP block injection, peak blood local anesthetic level after injection, the effect of spine movement (i.e., gliding movement of erector spinae muscle on the transverse processes) on neural blockade, and the consistency of this block technique. Also, most case reports on surgical patients did not report the onset, progression or resolution of ESP blockade or the extent of sensory and sympathetic blockade. From a clinical perspective, it would be very helpful to determine the extent and duration of clinical neural blockade following an ESP injection with different local anesthetic doses and such detailed examination is possible only in a carefully conducted volunteer study.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 (normal healthy) volunteers
* 18 - 50 years of age
* 60- 100 kg weight
* English speaking
* female volunteers of childbearing potential will be required to provide a negative pregnancy test before being allowed to participate, females of child bearing potential must be willing to use medically acceptable birth control methods for a minimum of 2 weeks following the nerve block.

Exclusion Criteria:

* weight < 60 kg (limited by the maximum lidocaine dose 7 mg/kg)
* medical disorders (including bleeding disorders)
* any recreational drug use
* allergy to local anesthetic (lidocaine, bupivacaine, ropivacaine)
* contraindication to regional anesthetic block
* inability to provide informed consent
* baseline abnormality of chest, abdominal and back sensation
* pregnancy / breast feeding
* individuals with mental health disorders (for example bipolar disorder or depression).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
the duration of sensory blockade Sensation to Pinprick of thoracic ventral rami | up to 10 hours
  duration of ESP block Sensation to Pinprick
the duration of sensory blockade Sensation to Pinprick of thoracic dorsal rami | up to 10 hours
  duration of ESP block Sensation to Pinprick
the duration of sensory blockade Sensation to temperature of thoracic ventral rami | up to 10 hours
  duration of ESP block Sensation to different temperature
the duration of sensory blockade Sensation to temperature of thoracic dorsal rami | up to 10 hours
  duration of ESP block Sensation to different temperature

SECONDARY OUTCOMES:
To evaluate the onset of pinprick blockade of an ESP block injection | up to 2 hours
  onset of ESP block on pinprick
To evaluate the onset of temperature blockade of an ESP block | up to 2 hours
  onset of ESP block on temperature
To evaluate the regression of pinprick blockade of an ESP block injection | post-block 2-10 hours
  regression of the ESP block on pinprick
To evaluate the regression of temperature blockade of an ESP block injection | post-block 2-10 hours
  regression of the ESP block on Skin Conductance
To evaluate the success of blockade on Skin Conductance of an ESP block injection | 0-2 hours
  post-block success of blockade on Skin Conductance
To evaluate the onset of blockade on Skin Conductance of an ESP block injection | post-block 0-2 hours
  the onset of blockade on Skin Conductance
To evaluate the regression of blockade on Skin Conductance of an ESP block injection | post-block 2-10hours
  the regression of blockade on Skin Conductance

CONTACTS AND LOCATIONS:
Overall Officials: Ki Jinn Chin, MBBS, MMed,FRCPC, Principal Investigator — UHN
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD with other researchers